CLINICAL TRIAL: NCT06774144
Title: Rezafungin Prophylaxis in Liver Transplant at High Risk for Invasive Fungal Infection
Brief Title: Rezafungin Prophylaxis in Liver Transplant
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Fernanda P Silveira, MD, MS (Other)
Collaborators: Melinta Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Fernanda P Silveira, MD, MS, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY24080165
Record Dates: First submitted 2024-12-18; First posted 2025-01-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Liver Transplant Infection; Fungal Infection
Keywords: rezafungin; liver transplant; prophylaxis
MeSH Terms: conditions — Mycoses | interventions — Rezafungin; Fluconazole; Voriconazole

STUDY DESIGN:
Intervention Model Description: Interventional, open-label, single center study with concurrent and historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prospective Intervention Cohort (Experimental): Rezafungin 400 mg IV once within 24 hours of liver transplant, followed by 200 mg IV once weekly for a total duration of 4 weeks
  Interventions: Drug: Rezafungin
- Prospective Control Cohort (Active Comparator): Patients who receive fluconazole/voriconazole or no antifungal prophylaxis as part of UPMC's risk-based antifungal prophylaxis standard of care after liver transplant
  Interventions: Drug: Standard of care antifungal prophylaxis
- Historical Control Group (Active Comparator): Patients at risk for IFI who received fluconazole/voriconazole for antifungal prophylaxis after liver transplant in the two years preceding the study
  Interventions: Drug: Standard of care antifungal prophylaxis

INTERVENTIONS:
Drug: Rezafungin — Rezafungin 400 mg IV once within 24 hours of liver transplant, followed by 200 mg IV weekly for 4 weeks.
  Arms: Prospective Intervention Cohort
Drug: Standard of care antifungal prophylaxis — UPMC uses a tiered approach to antifungal prophylaxis, based on risk factors for IFI. Fluconazole is used for recipients with risk factors for yeast infections: choledochojejunostomy, prolonged transplant time, receipt of >40 units of blood products within 24 hours of transplant, and Candida colonization or infection within 3 months prior to transplant. Voriconazole is used for recipients with risk factors for mould infections: re-transplantation, renal failure requiring renal replacement therapy, fulminant hepatic failure as indication for transplant, intra-abdominal/thoracic re-exploration within the first month after transplant. No prophylaxis is given if there are no risk factors for yeast or mould infections.
  Other Names: Fluconazole, voriconazole, or no prophylaxis
  Arms: Historical Control Group; Prospective Control Cohort

SUMMARY:
This is an interventional study to evaluate the efficacy of rezafungin, a new echinocandin, for the prevention of invasive fungal infections (IFIs) after liver transplantation. Patients who receive rezafungin will be compared to a similar group of patients who underwent liver transplantation in the preceding two years for the incidence of IFIs.

DETAILED DESCRIPTION:
This is a single arm interventional study of consecutive liver transplant recipients who have consented to this rezafungin prophylaxis study. The outcome will be compared with that of similar group of patients not enrolled in the study and those who underwent liver transplant in the preceding two years (historical controls). Propensity score matching will be used to select retrospective cohort.

There will be 3 groups:

1. Study group (prospective intervention cohort): Rezafungin (180 patients)
2. Prospective control group (prospective control cohort): Patients who receive fluconazole/voriconazole or no antifungal prophylaxis as part of UPMC's tiered antifungal prophylaxis standard of care (20 patients: 10 who receive fluconazole/voriconazole and 10 who do not receive fluconazole/voriconazole)
3. Historical control group (retrospective control cohort): Patients at risk for IFI who received fluconazole/voriconazole (tier approach) in the two years preceding this study (180 patients)

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipient
* 18 years of age or older
* ≥1 risk factor(s) for IFI: living donor transplant, retransplantation, complicated operations (based on duration of transplant and number of blood products required in the peri-transplant period), choledochojejunostomy anastomosis, or peri-operative Candida colonization, recent Candida infection, renal replacement therapy post-transplant, and reoperation within the first 90 days of transplant.

Exclusion Criteria:

* Participants who are perceived not to survive past 7 days after transplant
* Participants who elect not to participate in the prospective trial
* Participants who had active candidiasis at the time of transplant
* Participants with a history of allergy to an echinocandin
* Participants who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of proven and probable IFIs | 90 days post-transplant
  Incidence of proven and probable IFIs within 90 days post-transplant
Incidence of proven and probable breakthrough IFI | While receiving rezafungin, voriconazole, or fluconazole
  Incidence of breakthrough IFI while on specific antifungal prophylaxis

SECONDARY OUTCOMES:
Fungal-free survival | 90 days and 6 months post-transplant
  Number of participants without fungal infection
Fungal colonization | 90 days and 6 months post-transplant
  Number of participants with presence or growth of fungi without it causing active infection or disease
Graft rejection | 90 days and 6 months post-transplant
  Number of participants with liver allograft acute rejection
Graft loss | 90 days 6 months post-transplant
  Number of participants with failure of the liver allograft to function adequately or to remain viable
All-cause mortality | 90 days 6 months post-transplant
  Number of participants who die
Number of participants with premature discontinuation of prophylaxis | 90 days post-transplant
  Number of patients who experience an adverse event requiring premature discontinuation of antifungal prophylaxis
Overall incidence of development of antifungal resistance | Within 6 months of transplant
  Antifungal resistance of breakthrough fungal organisms or fungal organisms recovered within the first 6 months of transplant for patients who received rezafungin

OTHER OUTCOMES:
Pharmakokinectics (PK) of rezafungin | Up to 4 weeks post-transplant
  Pharmacokinetics of rezafungin while in ICU to assess the PK during the peri-transplant period
Stool microbiota composition | Within 6 months post-transplant
  Stool microbiota and fecal Candida constituent and susceptibility profile in response to rezafungin

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data outside of our investigative team and collaborators. Aggregate data will be shared in publications as appropriate.